CLINICAL TRIAL: NCT07072013
Title: An Indirect Treatment Comparison of the Effectiveness of Ribociclib Combined With Non-steroidal Aromatase Inhibitors vs. Tamoxifen for the Adjuvant Treatment of Premenopausal Women With Hormon Receptor-positive, HER2-negative Early Breast Cancer (IRINA)
Brief Title: An Indirect Treatment Comparison of the Effectiveness of Ribociclib Combined With Non-steroidal Aromatase Inhibitors vs. Tamoxifen for the Adjuvant Treatment of Premenopausal Women With Hormon Receptor-positive, HER2-negative Early Breast Cancer
Acronym: IRINA
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ADE10
Record Dates: First submitted 2025-07-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Ribociclib,; early breast cancer,; indirect treatment comparison,; tamoxifen,; premenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- tamoxifen±OFS external control arm: data were retrieved from the CLEAR-B study, provided by Institut für Frauengesundheit GmbH, Erlangen
  Interventions: Other: ribociclib
- Ribociclib+NSAI+OFS arm: Ribociclib+NSAI+OFS data for premenopausal women were sourced from NATALEE trial data
  Interventions: Other: ribociclib

INTERVENTIONS:
Other: ribociclib — This is an observational study. There is no treatment allocation. The decision to initiate ribociclib was based solely on clinical judgement.

SUMMARY:
The purpose of this indirect treatment comparison (ITC) was to generate comparative evidence on the effectiveness and safety in premenopausal women of ribociclib+Non-steroidal Aromatase Inhibitor (NSAI)+Ovarian Function Suppression (OFS) investigated in the global NATALEE trial (CLEE011O12301C, NCT 03701334) vs. tamoxifen±OFS using patients treated in German routine care as external control

DETAILED DESCRIPTION:
Data of premenopausal Early Breast Cancer (EBC) patients treated with tamoxifen±OFS in German routine care were used as external control for a patient-level adjusted ITC of ribociclib+NSAI+OFS vs. tamoxifen±OFS. The ribociclib+NSAI+OFS arm utilized data of premenopausal women in the NATALEE clinical trial. The tamoxifen±OFS arm as the external control used a subset of data collected in the CLEAR-B project (NCT05870813).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between 18 and 60 years
* HR-positive, HER2-negative EBC without distant metastases
* Patients must belong to one of the following categories according to the American Joint Committee on Cancer (AJCC):

  * Anatomic Stage Group III,
  * Anatomic Stage Group IIB,
  * Anatomic Stage Group IIA that it either:

    * N1,
    * N0 with the following criteria:
* Grade 3
* Grade 2, with any of the following criteria:

  * Ki67 ≥ 20 % or
  * Oncotype DX Breast Recurrence Score ≥ 26 or
  * Prosigna/PAM50 categorized as high risk or
  * MammaPrint categorized as high risk or
  * EndoPredict EPclin Risk Score categorized as high risk.
  * Patients with Cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor treatment other than ribociclib+NSAI+OFS were excluded
  * Patients in a bad general condition [Eastern Cooperative Oncology Group (ECOG) Status > 1] or with a limited life expectancy < 5 years were excluded

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: premenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 1937 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (iDFS) | 96 months
  Invasive Disease-Free Survival (iDFS) is defined as the time (in months) from the reference date to the date of the first contributing event and is censored otherwise.
  Contributing events according to the Standardized Definitions for Efficacy End Points (in Adjuvant Breast Cancer Trials) (STEEP) are
  * invasive ipsilateral breast tumor recurrence,
  * local/regional invasive recurrence,
  * distant recurrence,
  * death from BC,
  * death from non-BC cause,
  * death from unknown cause,
  * invasive contralateral BC,
  * or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin, or new in situ carcinomas of any site).
Distant Disease-Free Survival (dDFS) | 96 months
  Distant Disease-Free Survival (dDFS) is defined as the time (in months) from the reference date to the date of first contributing event. Contributing events according to the STEEP criteria are:
  * distant recurrence
  * death from BC
  * death from a non-BC cause
  * death from an unknown cause or
  * a second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin, or new in situ carcinomas of any site).
Recurrence-Free Survival (RFS) | 96 months
  Recurrence-Free Survival (RFS) is defined as the time (in months) from the reference date to the date of the first contributing event and censored otherwise. Contributing events according to STEEP are
  * invasive ipsilateral breast tumor recurrence,
  * local/regional invasive recurrence,
  * distant recurrence,
  * death from BC,
  * death from a non-BC cause,
  * death from an unknown cause.
Overall Survival (OS) | 96 months
  Overall survival (OS) is defined as the time (in months) from the reference date to the date of death from any cause. Time for censored patients is defined as the time from the reference date to last contact date.
Treatment Terminations (TT) | 96 months
  For the ribociclib+NSAI+OFS arm, Treatment Termination (TT) is defined as permanent treatment termination of treatment.
  For the tamoxifen±OFS arm, TT is defined as permanent termination of adjuvant tamoxifen.
Treatment Terminations due to Toxicity (TT_Tox) | 96 months
  For the ribociclib+NSAI+OFS arm, Treatment Termination due to Toxicity (TT_Tox) is defined as permanent treatment termination due to toxicity within three years of beginning ribociclib.
  For the tamoxifen±OFS arm, TT_Tox is defined as permanent treatment termination of adjuvant tamoxifen due to toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis investigative site, München, Germany

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com